CLINICAL TRIAL: NCT01787240
Title: Neurobiological Bases of Placebo Response in Major Depressive Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Cristina Cusin, MD, Instructor HMS, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012P001241
Record Dates: First submitted 2013-01-16; First posted 2013-02-08 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): After a screening visit, the patient will undergo a baseline assessment and will be randomized to escitalopram 10mg or placebo.
  Interventions: Drug: Placebo
- Escitalopram 10mg (Experimental): After a screening visit, the patient will undergo a baseline assessment and will be randomized to escitalopram 10mg or placebo.
  Interventions: Drug: Escitalopram 10mg

INTERVENTIONS:
Drug: Escitalopram 10mg
  Other Names: Lexapro
  Arms: Escitalopram 10mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
We are doing this research study to find out if people who get better while taking a specific kind of antidepressant medication (a selective serotonin reuptake inhibitor, or SSRI) and people who get better while taking placebo (an inactive substance) have similar chemicals in their brains. Some participants may complete a procedure called Acute Tryptophan Depletion (ATD), which is a way to study the role of serotonin in depression. Some participants may also undergo a magnetic resonance-positron emission tomography (MR-PET) scan.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for Major Depressive Disorder
* Written informed consent
* Men or women aged 18-60 years old
* A score of 18 or greater on the HAMD-28
* Patient must continue to meet criteria for current MDD at baseline. Patients must have Clinical Global Impression Improvement (CGI) scores ≥ 3 (i.e. minimally improved or less) from the screen to the baseline visit
* Agreeing to, and eligible for all procedures (only patients 18-45 will be eligible for MR-PET study)

Exclusion Criteria:

* Pregnant women or women of child bearing potential not using a medically accepted means of contraception
* Patients who are a serious suicide or homicide risk
* Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease, uncontrolled seizure disorder
* The following DSM-IV diagnoses: a) organic mental disorders b) substance use disorders, including alcohol, active within the last year; c) schizophrenia; d) delusional disorder; e) psychotic disorders not elsewhere classified; f) bipolar disorder; g) acute bereavement; h) borderline or antisocial personality disorder i) current primary diagnoses of panic disorder, social phobia, GAD, or OCD (disorders that present as chief complaint and/or have their onset preceding the onset of MDD), l) Patients with mood congruent or mood incongruent psychotic features
* Currently taking any of the following exclusionary medications: antipsychotics, anticonvulsants, mood stabilizers, stimulants, antidepressants, potential antidepressant augmenting agents (e.g., T3, SAMe, St. John's Wort, lithium, buspirone, Omega 3 fatty acids). If it is determined that it is safe to discontinue a medication, the patient will be required to wait a period equivalent to at least 5 half lives of the drug before the screening
* Patients who have taken an investigational psychotropic drug within the last year
* Patients who have not responded to one or more antidepressant trials of adequate doses (e.g., fluoxetine 40 mg/day or higher) and duration (e.g., for six weeks or more) over the past five years, as defined by the MGH-ATRQ
* History of inadequate response or poor tolerability to citalopram or escitalopram
* Any concomitant form of psychotherapy (depression-focused)
* Receiving or have received during the index episode Vagal nerve stimulation, ECT or rTMS, or other somatic antidepressant treatments
* Any reason not listed, determined by the site PI or study clinician, constituting good clinical practice and making participation in the study hazardous
* Contraindications to fMRI scanning and MR-PET scanning (including presence of a cardiac pacemaker or pacemaker wires, metallic particles in the body, vascular clips in the head or previous neurosurgery, prosthetic heart valves, claustrophobia)
* MR-PET-specific exclusion criteria: Patients who are younger than 18 or older than 45 years of age

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Cusin, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Depression Clinical and Research Program, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: After a screening visit, the patient will undergo a baseline assessment and will be randomized to escitalopram 10mg or placebo.
  Placebo
- Escitalopram 10mg: After a screening visit, the patient will undergo a baseline assessment and will be randomized to escitalopram 10mg or placebo.
  Escitalopram 10mg
Period: Overall Study
Arm/Group | Placebo | Escitalopram 10mg
Started | 15 | 5
Completed | 10 | 4
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Escitalopram 10mg | Total
Number analyzed (Participants) | 15 | 5 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 5 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.6 (14.10) | 33 (11.64) | 32.7 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 8 | 2 | 10
Region of Enrollment [Number; unit: participants]
  United States | 15 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Feasibility
Description: We will measure the percentage of screened eligible patients who agree to be randomized. Participants were assessed for this Outcome Measure before randomization.This would occur at the first study visit (screening).
Time Frame: This would occur at the first study visit (screening).
Measure: Number; unit: percent of eligible patients
Groups:
- Eligible Patients: Number of patients who were screened and were determined to be eligible for the study.
Arm/Group | Eligible Patients
Number analyzed (Participants) | 21
percent of eligible patients | 95.2

2. Secondary Outcome: Effects of Acute Tryptophan Depletion on Mood
Description: We will examine differences in scores on the the HAMD-28 before and after acute tryptophan depletion. Changes in these parameters will be compared between placebo responders and drug responders using unpaired two-tailed t-tests.
  The HAMD-28 measures depression severity, and has a minimum value of 0 and a maximum value of 81 units on a scale, where higher scores indicate more severe depression.
  A negative change value refers to a decrease in HAM D score.
Time Frame: Baseline, Visit 10 (after 9 weeks in study)
Population: Participants assigned to take either active drug or placebo who did not respond by the end of phase 1 (Week 5 of study treatment) continued onto phase 2.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Phase 2 Placebo: Participants assigned to take placebo who did not respond by the end of phase 1 (Week 5 of study treatment) continued onto phase 2.
- Phase 2 Active: Participants assigned to take active drug who did not respond by the end of phase 1 (Week 5 of study treatment) continued onto phase 2.
Arm/Group | Phase 2 Placebo | Phase 2 Active
Number analyzed (Participants) | 6 | 3
units on a scale | -6.0 (6.4) | -13.0 (12.1)

3. Secondary Outcome: Effects of Acute Tryptophan Depletion on Mood
Description: as for outcome 2
Time Frame: Baseline, Visit 5 (4 weeks into study)
Population: Patients who were randomized to take placebo or active drug
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Escitalopram 10mg
Number analyzed (Participants) | 12 | 4
units on a scale | -6.4 (8.5) | -8.8 (6.3)

4. Other Pre Specified Outcome: Effects of Acute Tryptophan Depletion on Serotonin Binding
Description: We will examine percentage changes in serotonin binding potential before and after acute tryptophan depletion within each region of interest. We will examine differences in serotonin binding potential between placebo responders and drug responders using a paired two-tailed t-test.
  Data were not collected
Time Frame: Visit 5 (after 4 weeks in study) or Visit 10 (after 9 weeks in study)
Population: Data were not collected
Arm/Group | Placebo | Escitalopram 10mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse event data were collected over the duration of the study, which lasted 2 years and 6 months.
Arm/Group | Placebo | Escitalopram 10mg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/5
Serious Adverse Events (participants affected / at risk) | 4/15 | 2/5
Other Adverse Events (participants affected / at risk) | 12/15 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Escitalopram 10mg (N=5)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Pancreatitis/Influenza (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Escitalopram 10mg (N=5)
Headache (Nervous system disorders) | 3 (5) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (2)
Gas/irregular Bowels (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anxiety attack (Psychiatric disorders) | 3 (3) | 0 (0)
Sleep paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Nervous system disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Chest pain/pressure (Cardiac disorders) | 1 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 0 (0)
Acid reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 2 (2) | 0 (0)
Memory issues (Psychiatric disorders) | 1 (1) | 0 (0)
Fatigue (Nervous system disorders) | 1 (2) | 0 (0)
Emotional lability (Psychiatric disorders) | 1 (1) | 0 (0)
Dry mouth (General disorders) | 1 (1) | 0 (0)
Heart palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Cold/sinus infection (Infections and infestations) | 1 (1) | 0 (0)
Bloated (Gastrointestinal disorders) | 1 (2) | 0 (0)
Sexual Interest/Libido (Psychiatric disorders) | 1 (5) | 0 (0)
Shoulder pain/numbness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No